CLINICAL TRIAL: NCT01578980
Title: Outpatient Control-to-Range: System and Monitoring Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); University of California, Santa Barbara (Other)
Responsible Party: Principal Investigator, Boris Kovatchev, PhD, Professor, Director of Center for Diabetes Technology, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16130
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Results first posted 2014-08-25 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-08

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Artificial Pancreas; Type 1 Diabetes Mellitus; Control-to-Range; Closed-Loop Control; Continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Outpatient Control-to-Range (Experimental): Outpatient Control-to-Range: Testing system connectivity
  Interventions: Device: Outpatient Control-to-Range

INTERVENTIONS:
Device: Outpatient Control-to-Range — Subjects will spend two nights (~42 hours) in a local hotel during which the AP Platform will be remotely monitored in an adjacent hotel room for validation that remote system monitoring can successfully occur.
  Other Names: Ambulatory Artificial Pancreas

SUMMARY:
A single arm, single treatment study is proposed to assess the feasibility of the AP Platform (cell phone + Control to Range system) outside of a hospital based clinical research center.

DETAILED DESCRIPTION:
Automated closed-loop control (CLC) of blood glucose, known as "artificial pancreas" (AP) can have tremendous impact on the health and lives of people with type 1 diabetes (T1DM). This inter-institutional and international research team has been on the forefront of CLC developments since the beginning of the Juvenile Diabetes Research Foundation (JDRF) Artificial Pancreas initiative in 2006. Thus far, the investigators have conducted three closed-loop control clinical trials (totaling 60 subjects with T1DM), which demonstrated significantly more time in an acceptable "target" blood glucose range during CLC, and significantly fewer hypoglycemic events during CLC compared to open loop. The overall objective is to sequentially test, validate, obtain regulatory approval for, and deploy at home, a closed-loop Control-to-Range (CTR) system comprised of two algorithmic components: a Safety Supervision Module (SSM) and a Hypoglycemia Mitigation Module (HMM). The SSM will monitor the safety of the subject's continuous subcutaneous insulin infusion pump (CSII) to prevent hypoglycemia and will also monitor the integrity of continuous glucose monitor (CGM) data for signal sensor deviations or loss of sensitivity. The HMM will be responsible for the optimal regulation of postprandial hyperglycemic excursions through correction boluses.

This study will test the ability of AP Platform to (1) run CTR in an outpatient setting, and (2) be remotely monitored. Specifically, this study involves studying adults with T1DM who are experienced insulin pump users. Subjects will spend two nights (~42 hours) in a local hotel, during which the AP Platform will be remotely monitored in an adjacent hotel room for validation that remote system monitoring can successfully occur. During the study, study subjects will be responsible for operating the CTR system with nursing and technicians available for additional support. A study physician and senior engineer will be on call.

Five subjects each will be enrolled at University of Virginia and the University of California, Santa Barbara.

ELIGIBILITY:
INCLUSION CRITERIA

1. ≥21 and <65 years old
2. Clinical diagnosis of type 1 diabetes mellitus:

   * Criteria for documented hyperglycemia (at least 1 criterion must be met):

     * Fasting glucose ≥126 mg/dL - confirmed
     * Two-hour Oral Glucose Tolerance Test (OGTT) glucose ≥200 mg/dL - confirmed
     * HbA1c ≥6.5% documented by history - confirmed
     * Random glucose ≥200 mg/dL with symptoms
     * No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with diabetes
   * Criteria for requiring insulin at diagnosis (at least 1 criterion must be met):

     * Participant required insulin at diagnosis and continually thereafter
     * Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually
     * Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually
3. Use of an insulin pump to treat his/her diabetes for at least 1 year
4. Actively using an insulin pump with bolus calculator feature including predefined parameters for carbohydrate ratio, insulin sensitivity factor, target blood glucose (BG) and active insulin.
5. HbA1c between 6.0% - 9.0% as measured with DCA2000 or equivalent device
6. Not currently known to be pregnant, breast feeding, or intending to become pregnant (females)
7. Demonstration of proper mental status and cognition for the study
8. Willingness to avoid consumption of acetaminophen-containing products during the study interventions
9. If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, have stability on the medication for at least 2 months prior to enrollment in the study

EXCLUSION CRITERIA

1. Diabetic ketoacidosis within the 6 months prior to enrollment
2. Severe hypoglycemia resulting in seizure, loss of consciousness, or 3rd party assistance in the 12 months prior to enrollment
3. Subject reports that he/she has hypoglycemia unawareness with severe low blood sugars (e.g. <50 mg/dL without symptoms)
4. Pregnancy; breast feeding, or intention of becoming pregnant
5. Uncontrolled arterial hypertension (diastolic blood pressure >90 mmHg and/or systolic blood pressure >160 mmHg)
6. Conditions which may increase the risk of hypoglycemia such as any cardiac disorder/arrhythmia, uncontrolled coronary artery disease during the previous year (e.g. history of myocardial infarction, acute coronary syndrome, therapeutic coronary intervention, coronary bypass or stenting procedure, stable or unstable angina, episode of chest pain of cardiac etiology with documented EKG changes, or positive stress test or catheterization with coronary blockages >50%), congestive heart failure, history of cerebrovascular event, seizure disorder, syncope, adrenal insufficiency, neurologic disease or atrial fibrillation
7. Hematocrit <40% (males) and <35% (females)
8. History of a systemic or deep tissue infection with methicillin-resistant staph aureus or Candida albicans
9. Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the CGM (implantable cardioverter-defibrillator, electronic pacemaker, neurostimulator, intrathecal pump, and cochlear implants)
10. Anticoagulant therapy other than aspirin
11. Oral steroids
12. Medical condition requiring use of an acetaminophen-containing medication that cannot be withheld for the study admissions.
13. Psychiatric disorders that would interfere with study tasks (e.g. inpatient psychiatric treatment within 6 months prior to enrollment)
14. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
15. Known current or recent alcohol or drug abuse
16. Medical conditions that would make operating a CGM, cell phone, or insulin pump difficult (e.g. blindness, severe arthritis, immobility)
17. Any skin condition that prevents sensor or pump placement on the abdomen or arm (e.g. bad sunburn, pre-existing dermatitis, intertrigo, psoriasis, extensive scarring, cellulitis)
18. Impaired hepatic function measured as alanine aminotransferase or aspartate aminotransferase ≥three times the upper reference limit
19. Impaired renal function measured as creatinine >1.2 times above the upper limit of normal
20. Uncontrolled microvascular (diabetic) complications (other than diabetic non-proliferative retinopathy), such as current proliferative diabetic retinopathy, known diabetic nephropathy (other than microalbuminuria with normal creatinine) or neuropathy requiring treatment
21. Active gastroparesis requiring current medical therapy
22. If taking antihypertensive, thyroid, anti-depressant or lipid lowering medication, lack of stability on the medication for the past 2 months prior to enrollment in the study
23. Uncontrolled thyroid disease
24. Known bleeding diathesis or dyscrasia
25. Known allergy to medical adhesives, components of the insulin pump insertion set or continuous glucose monitor sensor
26. Active enrollment in another clinical trial
27. Unwillingness to withhold dietary supplements two weeks prior to admission and for the duration of the study participation
28. Use of anti-diabetic agents other than CSII including long-acting insulin, intermediate-acting insulin, metformin, sulfonylureas, meglitinides, thiazolidinediones, DPP-IV inhibitors, glucagon-like peptide 1 agonists, and alpha-glucosidase inhibitors
29. Subjects with basal rates less than 0.05.

RESTRICTIONS ON USE OF OTHER DRUGS OR TREATMENTS.

1. Use of anti-diabetic agents other than CSII including long-acting insulin, intermediate-acting insulin, metformin, sulfonylureas, meglitinides, thiazolidinediones, DPP-IV inhibitors, glucagon-like peptide 1 agonists, and alpha-glucosidase inhibitors.
2. Oral steroids are excluded
3. Anticoagulant therapy other than aspirin is excluded
4. Acetaminophen will not be allowed while the continuous glucose monitor is in use
5. Dietary supplements will be withheld two weeks prior to admission and for the duration of study participation
6. Medications that block symptoms of hypoglycemia, including but not limited to beta blockers

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris P. Kovatchev, Ph.D., Study Chair — University of Virginia
Locations (2):
- United States (2):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Result] Kovatchev BP, Renard E, Cobelli C, Zisser HC, Keith-Hynes P, Anderson SM, Brown SA, Chernavvsky DR, Breton MD, Farret A, Pelletier MJ, Place J, Bruttomesso D, Del Favero S, Visentin R, Filippi A, Scotton R, Avogaro A, Doyle FJ 3rd. Feasibility of outpatient fully integrated closed-loop control: first studies of wearable artificial pancreas. Diabetes Care. 2013 Jul;36(7):1851-8. doi: 10.2337/dc12-1965. PMID 23801798

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Outpatient Control-to-Range
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Outpatient Control-to-Range
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 10
  France | 5
  Italy | 5
HbA1c 6-9% [Number; unit: participants] | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent Time of Active CTR
Description: The main endpoint will be the percent time with all expected data from CGM, pump and patient manual inputs that should be available on Artificial Pancreas platform and monitoring stations. To be considered as successful, this percent time will have to reach more than 80% of total time of investigation for the entire arm.
Time Frame: 42 hours
Population: The three pilot subjects (one for each country) were not included in the analysis.
Measure: Number; unit: percentage of time of active CTR
Groups:
- Outpatient Control-to-Range: Outpatient Control-to-Range: Testing system connectivity
  Outpatient Control-to-Range: Subjects will spend two nights (~42 hours) in a local hotel during which the AP Platform will be remotely monitored in an adjacent hotel room for validation that remote system monitoring can successfully occur.
  42 hours total: 14 hours in open-loop 28 hours in closed-loop
Arm/Group | Outpatient Control-to-Range
Number analyzed (Participants) | 17
percentage of time of active CTR | 98

2. Secondary Outcome: Frequency of Unplanned System Resets or Restarts
Description: Frequency of unplanned system resets or restarts
  Secondary endpoints include the estimation of the failure rates of system components, frequency analysis of lost or inaccurate CGM records, and percent time of active CTR. The failure/missing data records will be compared to failure/missing data records from our past in-clinic studies.
Time Frame: 42 hours
Population: The three pilot subjects (one for each country) were not included in the analysis.
Measure: Number; unit: events per 24 hours
Arm/Group | Outpatient Control-to-Range
Number analyzed (Participants) | 17
events per 24 hours
  Viliv S5 tablet (n=7) | 2.89
  Galaxy Nexus phone (n=10) | 0.58

ADVERSE EVENTS:
Time Frame: 42 hours
Arm/Group | Outpatient Control-to-Range
Serious Adverse Events (participants affected / at risk) | 9/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Outpatient Control-to-Range (N=20)
Hypoglycemia (Endocrine disorders) | 6 (6) — Hypoglycemia <60 mg/dL requiring carbohydrate treatment
Staff Initiated System Shut-dowm (Endocrine disorders) | 3 (3) — Hyperglycemia due to site failure or tube occlusion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes